CLINICAL TRIAL: NCT07270523
Title: Therapeutic Monitoring of Beta-lactams in Critically Ill Patients With Sepsis: OPTIBETA Clinical Trial Protocol
Brief Title: Therapeutic Monitoring of Beta-lactams in Critically Ill Patients With Sepsis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Complexo Hospitalario Universitario de A Coruña (Other)
Collaborators: Hospital Clínico Universitario de Santiago de Compostela (Unknown)
Responsible Party: Principal Investigator, Manuel Ángel Gómez-Ríos, Anesthesiologist, Complexo Hospitalario Universitario de A Coruña
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPTIBETA
Record Dates: First submitted 2025-11-14; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Bacterial Sepsis
Keywords: betalactam; therapeutic drug monitoring; sepsis; clinical cure; microbiological cure
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: OPTIBETA is a pragmatic, randomized, controlled, low-intervention, hospital-based clinical trial. Patients will be randomly assigned in a 1:1 ratio to one of the following groups:
  * Intervention: individualized dosing of beta-lactam antibiotics guided by therapeutic drug monitoring (TDM) with adjustment according to pharmacokinetic/pharmacodynamic (PK/PD) targets.
  * Control: standard dosing based on clinical guidelines, without individualized adjustment.
  The study will be open-label, although the evaluators of clinical and microbiological outcomes will be blinded to treatment assignment in order to reduce observation bias.
Who Masked: Outcomes Assessor
Masking Description: The randomization sequence will be generated using independent software (randomization.com). Concealment will be ensured using opaque, sequentially numbered envelopes and an electronic case report form (eCRF) that is locked until assignment. Outcome assessors will remain blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (individualized dosing based on therapeutic monitoring) (Experimental): Patients will receive individualized dosing of beta-lactam antibiotics based on therapeutic monitoring. Total and free plasma concentrations will be determined 48 hours after the start of antibiotic therapy and subsequently every 4-5 days, or sooner if there is a significant clinical change. Dosage adjustments will be made to achieve the defined PK/PD targets:
  * Standard: ≥100% fT > MIC.
  * Infections caused by multidrug-resistant pathogens, increased renal clearance, or immunosuppression: ≥100% fT > 4×MIC.
  Concentrations will be interpreted in relation to the actual MIC of the identified pathogen or, failing that, to the ECOFF values defined by EUCAST.
  Interventions: Other: Individualized dosing of beta-lactam antibiotics based on therapeutic monitoring
- Control group (usual dosage): (No Intervention): Patients will receive the usual dosage of beta-lactam antibiotics following the recommendations of clinical guidelines and hospital protocols, without individualized adjustment based on MDT. Plasma samples will also be collected, but will be stored for deferred analysis at the end of the study, with no impact on clinical management.

INTERVENTIONS:
Other: Individualized dosing of beta-lactam antibiotics based on therapeutic monitoring — In the intervention group, plasma levels will be determined 48 hours after the start of antibiotic treatment and subsequently every 4-5 days, with a pharmacotherapeutic report and dosage adjustment within <24 hours. In the control group, samples will be stored at -80 °C and analyzed at the end of the study, with no impact on clinical practice.
  Plasma concentrations of beta-lactam antibiotics will be determined by high-performance liquid chromatography (HPLC) using validated commercial kits, which allow simultaneous quantification of several drugs in this group with reduced processing times and feasible implementation in hospital routine.
  Patients will be evaluated weekly until hospital discharge, death, or completion of antibiotic treatment. Clinical progression, inflammatory markers, emergence of resistance, adverse effects, and clinical and microbiological outcomes will be recorded.
  Arms: Intervention group (individualized dosing based on therapeutic monitoring)

SUMMARY:
Background: Sepsis is a leading cause of morbidity and mortality among critically ill patients and is associated with intensive use of β-lactam antibiotics. These drugs show time-dependent pharmacodynamics and high pharmacokinetic variability in this population, making it difficult to achieve therapeutic levels. Therapeutic drug monitoring (TDM) may optimize dosing, but its routine clinical implementation remains limited.

Objective: To evaluate whether individualized β-lactam dosing guided by TDM reduces time to full clinical recovery compared with standard dosing in critically ill patients with sepsis.

Methods: OPTIBETA is a pragmatic, randomized, controlled, open-label clinical trial to be conducted at a tertiary hospital in Spain. Adult patients (≥18 years) admitted to the intensive care unit or infectious diseases ward with sepsis will be included. Participants will be randomized 1:1 to either a TDM-guided dosing arm (dose adjustments according to PK/PD targets) or a standard dosing arm. Clinical, microbiological, and pharmacological outcomes will be collected. The primary endpoint is time to complete clinical cure. Secondary outcomes include overall survival, microbiological cure, ICU and hospital length of stay, adverse events, and achievement of PK/PD targets. The estimated sample size is 198 patients.

Expected results: We hypothesize that TDM-guided dosing will reduce time to clinical cure, improve overall outcomes, and decrease adverse events compared with standard dosing.

Conclusions: OPTIBETA will provide high-quality evidence on the role of β-lactam TDM in critically ill septic patients and may support its inclusion in antimicrobial stewardship programs.

DETAILED DESCRIPTION:
Sepsis is a global health problem of enormous magnitude, responsible for more than 48 million cases and 11 million deaths annually, accounting for around 20% of global mortality. Its prevalence is particularly high in critically ill patients, occurring in up to 40% of ICU admissions. In Spain, it causes more than 17,000 deaths per year, exceeding the mortality rate of some types of cancer. In addition to its clinical impact, sepsis entails a considerable economic burden, with direct costs estimated at between €20,000 and €30,000 per patient admitted to the ICU, to which must be added indirect costs arising from functional sequelae and loss of productivity. Early and appropriate antibiotic treatment is essential to improve prognosis, with beta-lactam antibiotics being the most widely used group due to their broad spectrum of action and safety profile. These drugs have time-dependent pharmacodynamics and high pharmacokinetic variability in septic patients, conditioned by factors such as multiple organ dysfunction, increased distribution volume, and renal hyperfiltration. These alterations make it difficult to achieve adequate therapeutic concentrations and can lead to both underdosing-associated with therapeutic failure and the development of resistance-and overdosing, with an increased risk of toxicity, especially neurological toxicity. These alterations make it difficult to achieve adequate therapeutic concentrations and can lead to both underdosing-associated with therapeutic failure and the development of resistance-and overdosing, with an increased risk of toxicity, especially neurological toxicity.

Therapeutic drug monitoring (TDM) applied to beta-lactam antibiotics allows for individualized dosage adjustment based on pharmacokinetic/pharmacodynamic (PK/PD) targets. Despite strong observational evidence supporting this strategy, its clinical implementation remains limited due to technical, organizational, and economic barriers, and the absence of pragmatic randomized clinical trials makes it difficult to establish its true impact on healthcare practice.

In this context, the OPTIBETA project hypothesizes that personalized dosing of beta-lactam antibiotics guided by MDT improves time to clinical cure compared to standard dosing in critically ill patients with sepsis. The primary objective of this trial is to evaluate the efficacy of individualized dosing based on MDT versus the conventional regimen in terms of reducing the time to complete clinical cure.

Hypothesis:

The administration of beta-lactam antibiotics adjusted to PK/PD targets in critically ill patients with sepsis based on plasma level determination improves clinical and microbiological cure compared to standard dosing.

Objectives:

The overall objective is to evaluate the efficacy and safety of personalized dosing of beta-lactam antibiotics based on TDM, compared to standard dosing, in critically ill patients with sepsis.

* Primary objective Evaluate whether individualized dosing of beta-lactam antibiotics based on pharmacokinetic monitoring and achievement of PK/PD targets is superior to standard dosing in terms of reducing the time to complete clinical cure (resolution of signs and symptoms of infection, functional recovery, baseline or improved SOFA score (≤2 points), and absence of need for new antibiotics).
* Secondary objectives

  * To evaluate the overall clinical efficacy of personalized dosing versus conventional dosing using variables such as: survival rate, clinical and microbiological cure rate, total length of hospital stay, number of days free of life-support therapies (vasopressors, renal replacement therapies, extracorporeal membrane oxygenation (ECMO)).
  * Analyze the emergence of antimicrobial resistance in both groups.
  * Compare the incidence of adverse effects (nephrotoxicity, hepatotoxicity, and neurotoxicity) between the personalized dosing group and the control group.
  * Determine the percentage of patients who achieve the established PK/PD targets: ≥100% fT > MIC or ≥100% fT > 4×MIC.
  * Study the influence of clinical variables (type of infection, microorganism involved, severity of clinical symptoms, etc.) on the probability of achieving PK/PD targets.
  * Evaluate the relationship between the total concentration and the free fraction of the antibiotic, and its impact on achieving the desired PK/PD parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Diagnosis of sepsis according to Sepsis-3 (SOFA ≥2).
* Initiation of treatment with beta-lactam antibiotics.
* Informed consent signed by the patient or their legal representative within the first 48 hours after the start of antibiotic therapy.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Known hypersensitivity to beta-lactams.
* Discontinuation of antibiotic treatment before the first TDM determination.
* Simultaneous participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Time to complete clinical cure | From the date of randomization to the date of clinical cure, assessed every 7 days and until the end of the study, an average of 3 years.
  The primary endpoint will be the time to complete clinical cure, defined as resolution of signs and symptoms of infection, functional recovery, baseline or improved SOFA score (≥2 points from baseline), and no need to initiate new antibiotic treatment.

SECONDARY OUTCOMES:
Time to microbiological cure (negative cultures). | From the date of randomization to the date of microbiological cure, assessed every 7 days and until the end of the study, an average of 3 years
  Time until microbiological cultures become negative
Overall survival (OS) | From the start date of treatment until the end of the study, an average of 3 years.
  Length of time that patients remain alive after start of treatment.
Length of hospital stay | From the date of randomization until the end of the study, an average of 3 years.
  Number of days the patient remains hospitalized
Number of days free of life support | From the date of randomization until the end of the study, an average of 3 years.
  Number of days free of life support (vasopressors, renal replacement therapy, extracorporeal membrane oxygenation).
Security | From the start date of treatment until the end of the study, an average of 3 years.
  Incidence of adverse effects related to beta-lactam antibiotics (nephrotoxicity, hepatotoxicity, and neurotoxicity).
Percentage of patients reaching established pharmacokinetics/pharmacodynamic (PK/PD) targets | From the date of randomization to the date of clinical cure, assessed every 4-5 days and until the end of the study, an average of 3 years.
  Percentage of patients out of the total number of patients included in the study who achieve the PK/PD objective in any of the measurements taken throughout the study, with this PK/PD objective being set at 100% fT > MIC or ≥100% fT > 4×MIC, depending on clinical profile.
Ratio between total and free concentrations of beta-lactam antibiotics. | From the date of randomization to the date of clinical cure, assessed every 4-5 days and until the end of the study, an average of 3 years.
  The ratio between the free beta-lactam concentration in the blood and the total concentration in each patient will be related, allowing relationships to be established between this ratio and the scope of the proposed PK/PD objective for that patient.
Identification of causative pathogens and their minimum inhibitory concentrations (MIC). | From the date of randomization until the end of the study, an average of 3 years.
Determination of the mechanism of antimicrobial resistance developed by the causative microorganism during treatment. | From the start date of treatment until the end of the study, an average of 3 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital of Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suarez D, Ferrer R, Artigas A, Azkarate I, Garnacho-Montero J, Goma G, Levy MM, Ruiz JC; Edusepsis Study Group. Cost-effectiveness of the Surviving Sepsis Campaign protocol for severe sepsis: a prospective nation-wide study in Spain. Intensive Care Med. 2011 Mar;37(3):444-52. doi: 10.1007/s00134-010-2102-3. Epub 2010 Dec 9. PMID 21152895
- [Background] Angus DC, van der Poll T. Severe sepsis and septic shock. N Engl J Med. 2013 Aug 29;369(9):840-51. doi: 10.1056/NEJMra1208623. No abstract available. PMID 23984731
- [Background] Sakr Y, Jaschinski U, Wittebole X, Szakmany T, Lipman J, Namendys-Silva SA, Martin-Loeches I, Leone M, Lupu MN, Vincent JL; ICON Investigators. Sepsis in Intensive Care Unit Patients: Worldwide Data From the Intensive Care over Nations Audit. Open Forum Infect Dis. 2018 Nov 19;5(12):ofy313. doi: 10.1093/ofid/ofy313. eCollection 2018 Dec. PMID 30555852
- [Background] Rudd KE, Johnson SC, Agesa KM, Shackelford KA, Tsoi D, Kievlan DR, Colombara DV, Ikuta KS, Kissoon N, Finfer S, Fleischmann-Struzek C, Machado FR, Reinhart KK, Rowan K, Seymour CW, Watson RS, West TE, Marinho F, Hay SI, Lozano R, Lopez AD, Angus DC, Murray CJL, Naghavi M. Global, regional, and national sepsis incidence and mortality, 1990-2017: analysis for the Global Burden of Disease Study. Lancet. 2020 Jan 18;395(10219):200-211. doi: 10.1016/S0140-6736(19)32989-7. PMID 31954465
- [Background] Perner A, Gordon AC, De Backer D, Dimopoulos G, Russell JA, Lipman J, Jensen JU, Myburgh J, Singer M, Bellomo R, Walsh T. Sepsis: frontiers in diagnosis, resuscitation and antibiotic therapy. Intensive Care Med. 2016 Dec;42(12):1958-1969. doi: 10.1007/s00134-016-4577-z. Epub 2016 Oct 1. PMID 27695884
- [Background] Reinhart K, Daniels R, Kissoon N, Machado FR, Schachter RD, Finfer S. Recognizing Sepsis as a Global Health Priority - A WHO Resolution. N Engl J Med. 2017 Aug 3;377(5):414-417. doi: 10.1056/NEJMp1707170. Epub 2017 Jun 28. No abstract available. PMID 28658587
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338